CLINICAL TRIAL: NCT05085613
Title: A Randomized Controlled Trial Testing the Efficacy of Humor and Framing in Messaging to Correct Misperceptions About COVID-19 Vaccines
Brief Title: Does Framing and Humor Improve the Effectiveness of Messages About COVID-19 Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00015120B
Record Dates: First submitted 2021-10-01; First posted 2021-10-20 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Beliefs

STUDY DESIGN:
Intervention Model Description: Model Description: Participants will be randomized to view one of four messages. The control message explains why people are hesitant to accept the FDA authorized COVID vaccines are safe and effective and how they are evaluated. Arm 2 additionally includes consequent framing regarding economic recovery (e.g. "If everyone gets vaccinated, we can keep schools, stores, and other businesses open so more Americans can keep working and supporting their families." With a picture of an "open for business" sign), arm 3 includes consequent framing regarding freedom to behave as one chooses (e.g. "Everyone getting vaccinated is the key to freedom! A vaccine can give us the freedom to hang out with friends, shop, and worship together again safely." With a picture of an American flag), and arm 4 includes humor (e.g. "Unfortunately, everyone getting vaccinated means leaving the house again.").
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vaccine Corrective Control (Active Comparator): A message that explains why people are hesitant to accept the FDA authorized COVID vaccines are safe and effective and how the vaccines are evaluated as safe and effective by FDA.
  Interventions: Behavioral: Corrective message framing and humor
- Vaccine corrective with economic recovery framing (Experimental): The content of the control message with the addition of the text, "If everyone gets vaccinated, we can keep schools, stores, and other businesses open so more Americans can keep working and supporting their families." The message will also include a picture of an "open for business" sign.
  Interventions: Behavioral: Corrective message framing and humor
- Vaccine corrective with freedom framing (Experimental): The content of the control message with the addition of the text, "Everyone getting vaccinated is the key to freedom! A vaccine can give us the freedom to hang out with friends, shop, and worship together again safely." The message will also include a picture of an American flag.
  Interventions: Behavioral: Corrective message framing and humor
- Vaccine corrective with humor (Experimental): The content of the control message with the addition of the text, "Unfortunately, everyone getting vaccinated means leaving the house again." The message will include a meme of a cat being pulled/rescued from a window with text boxes labeling the cat as "People at home working in sweatpants" and the rescuer as "COVID Vaccines."
  Interventions: Behavioral: Corrective message framing and humor

INTERVENTIONS:
Behavioral: Corrective message framing and humor — The main content of the messages will be the same. Experimental conditions (arms 2-4) will additionally include consequent framing as a result of getting vaccinated (e.g. economic recovery for arm 2 and freedom for arm 3) and humor for arm 4. Participants will be randomized to view one of the four messages.

SUMMARY:
This study seeks to assess the efficacy of educational messages to correct misperceptions. People hold a number of misperceptions that are relevant to public health, including misperceptions regarding COVID vaccines. Some people incorrectly think the COVID vaccines authorized by FDA are not safe or effective. These misperceptions can reduce adherence to public health recommendations and result in continued spread of COVID. This study will test if humor and different types of framing increase the efficacy of messages to correct misperceptions about FDA's authorized coronavirus vaccine safety and effectiveness. The frames tested will include: framing the vaccine as a way to boost economic recovery and framing the vaccine as a way to increase freedom to choose how to behave. The addition of humor will also be tested. Message efficacy will be measured via improved accuracy of beliefs after being exposed to the message. In other words, participants will be asked how safe and effective FDA authorized COVID vaccines are before seeing a message, then they will see a message about why the COVID vaccines are safe and effective, and then they will again be asked how safe and effective they think the vaccines are. This study will also assess the accuracy of inferential beliefs. This will be accomplished by asking participants questions about other vaccines that either are or are not authorized by FDA. If participants have understood the messages and updated their mental models of how FDA evaluates vaccines, they should be able to infer if other vaccines are safe and effective based on their FDA authorization status.

Hypotheses

H1: Participants who are exposed to A.) a message with humor, B.) a message with an economic recovery fame, or C.) a message with a freedom frame will be more likely to increase their agreement with the statement that the FDA will only authorize coronavirus vaccines that are safe and effective after message exposure than participants exposed to the control condition.

H2: Participants who are exposed to A.) a message with humor, B.) a message with an economic recovery fame, or C.) a message with a freedom frame will agree more strongly with the statement that the FDA approved flu vaccine is safe and effective after message exposure than participants exposed to the control condition.

H3. Participants who are exposed to A.) a message with humor, B.) a message with an economic recovery fame, or C.) a message with a freedom frame will agree more strongly with the statement that the ResVax vaccine, which was not approved by the FDA for the treatment of RSV, is a safe and effective after message exposure than participants exposed to the control condition.

H4. Participants who are exposed to A.) a message with humor, B.) a message with an economic recovery fame, or C.) a message with a freedom frame will be more likely to increase behavioral intentions to get an FDA authorized COVID vaccine after message exposure than participants exposed to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Are 21 years of age or older.
* Have not participated in the cognitive interview.
* Have not yet received a COVID vaccine.
* Are registered with MTurk in the United States.
* Have completed >= 5,000 HIITs within the MTurk system
* Have a HIIT approval rating of >= 97%
* Rate their agreement with the following statement as less than or equal to 50 out of 100: "To what extent do you agree with the following: "The FDA only authorizes COVID vaccines that are safe and effective."

Exclusion Criteria:

* Are younger than 21 years of age
* Participated in the cognitive interviews
* Have already received a COVID vaccine.
* Are not registered with MTurk in the US
* Have completed < 5,000 HIITS
* Have a HIIT approval rating of <97%
* Rate their agreement with the following statement as greater than 50 out of 100: "To what extent do you agree with the following: "The FDA only authorizes COVID vaccines that are safe and effective."

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Moran, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, deidentified participant data collected during the study may be shared. Upon request, we may also share the study protocol, survey, and informed consent form. Data will be made available upon request beginning 3 months following publication of the final article from this study, with no end date. Data will be made available for analyses deemed appropriate by the study PI. Proposals should be directed to mmoran22@jhu.edu. Data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 3 months following publication of the final article from this study, with no end date.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor
Started | 27 | 27 | 24 | 22
Completed | 27 | 27 | 24 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor | Total
Number analyzed (Participants) | 27 | 27 | 24 | 22 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (9.9) | 41.4 (11.9) | 43.3 (9.2) | 40.8 (9.7) | 41.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 10 | 9 | 42
  Male | 19 | 12 | 14 | 13 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 19 | 24 | 20 | 16 | 79
  Race/ethnicity: Racial/ethnic minority | 8 | 3 | 4 | 6 | 21
Political affiliation [Count of Participants; unit: Participants]
  Conservative | 11 | 18 | 16 | 13 | 58
  Liberal | 3 | 4 | 6 | 3 | 16
  Moderate | 13 | 5 | 2 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Accuracy of the Belief That FDA Authorized COVID-19 Vaccines Are Safe and Effective
Description: Assessed by change in response to the question To what extent do you agree or disagree with the following statement: The FDA has only authorized COVID vaccines that are safe and effective; with response options on a continuous scale from 0 "I do not agree at all" to 100, "I completely agree."
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Mean (Standard Deviation); unit: score on a 0-100 scale
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor
Number analyzed (Participants) | 27 | 27 | 24 | 22
score on a 0-100 scale | 20.1 (23.8) | 22.8 (24.0) | 24.2 (26.9) | 22.7 (24.1)
Statistical Analysis 1: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Economic Recovery Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.998, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF=6; Mean Difference (Final Values) = .6279928, 95% CI 2-sided [-9.463627 to 10.71961], Standard Error of Mean 4.150369 — Economic recovery condition - control
Statistical Analysis 2: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Freedom Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.725, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = 4.044194, 95% CI 2-sided [-6.416608 to 14.505], Standard Error of Mean 4.302202 — Freedom - control
Statistical Analysis 3: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Humor; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.980, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = -1.53656, 95% CI 2-sided [-12.25295 to 9.179834], Standard Error of Mean -1.53656 — Humor - control

2. Primary Outcome: Accuracy of Inferential Belief That the FDA Authorized Flu Vaccine is Safe and Effective
Description: Assessed by response to the question To what extent do you agree with the following: The FDA authorized flu vaccine is safe and effective.; with response options on a continuous scale from 0 "I do not agree at all" to 100, "I completely agree."
Time Frame: Up to 5 minutes after receiving the corrective message
Measure: Mean (Standard Deviation); unit: score on a 0-100 scale
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor
Number analyzed (Participants) | 27 | 27 | 24 | 22
score on a 0-100 scale | 37.074074 (33.546668) | 44.666667 (31.619128) | 49.583333 (35.808569) | 50.954545 (35.18993)
Statistical Analysis 1: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Economic Recovery Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.813, ANCOVA — Sidak's adjusted p-value for multiple comparisons; Df = 6; Mean Difference (Final Values) = 7.002255, 95% CI 2-sided [-14.39448 to 28.39899], Standard Error of Mean 8.801527 — Economic recovery condition - control
Statistical Analysis 2: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Freedom Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.268, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = 15.12214, 95% CI 2-sided [-6.938055 to 37.18234], Standard Error of Mean 9.07444 — Freedom - control
Statistical Analysis 3: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Humor; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.330, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = 14.4032, 95% CI 2-sided [-8.218891 to 37.0253], Standard Error of Mean 9.305576 — Humor - Control

3. Primary Outcome: Accuracy of Inferential Belief That RexVax is Safe and Effective
Description: Assessed by response to the question, The FDA recommended more testing of ResVax and did NOT authorize the vaccine because it did not prevent enough RSV infections.
  To what extent do you agree with the following: ResVax is safe and effective; with response options on a continuous scale from 0 "I do not agree at all" to 100, "I completely agree."
Time Frame: Up to 5 minutes after receiving the corrective message
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor
Number analyzed (Participants) | 27 | 27 | 24 | 22
units on a scale | 14.923077 (20.853629) | 14.24 (23.502269) | 12.47619 (17.28473) | 23.863636 (28.782097)
Statistical Analysis 1: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Economic Recovery Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.994, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 5; Mean Difference (Final Values) = -1.457003, 95% CI 2-sided [-16.98852 to 14.07451], Standard Error of Mean 6.380984 — Economic recovery - control
Statistical Analysis 2: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Freedom Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.998, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 5; Mean Difference (Final Values) = -1.097586, 95% CI 2-sided [-17.34491 to 15.14973], Standard Error of Mean 6.675066 — Freedom - control
Statistical Analysis 3: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Humor; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.447, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 5; Mean Difference (Final Values) = 8.926191, 95% CI 2-sided [-7.110771 to 24.96315], Standard Error of Mean 6.588643 — Humor - Control

4. Primary Outcome: Change in Intention to Get a COVID-19 Vaccine
Description: Assessed by change in response to the statement: I plan on getting an FDA authorized coronavirus vaccine; with response options on a continuous scale from 0 "I do not agree at all" to 100, "I completely agree."
Time Frame: Baseline and up to 5 minutes after receiving the corrective message
Measure: Mean (Standard Deviation); unit: score on a 0-100 scale
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor
Number analyzed (Participants) | 27 | 27 | 24 | 22
score on a 0-100 scale | 15.925926 (24.935187) | 9.4814815 (16.032108) | 9.625 (21.906546) | 12.863636 (20.2797)
Statistical Analysis 1: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Economic Recovery Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.113, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = -4.154612, 95% CI 2-sided [-8.985328 to .6761041], Standard Error of Mean 1.986723 — Economic recovery - control
Statistical Analysis 2: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Freedom Framing; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.473, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = -2.685896, 95% CI 2-sided [-7.66090 to 2.289114], Standard Error of Mean 2.046067 — Freedom - control
Statistical Analysis 3: Comparison: Vaccine Corrective Control vs Vaccine Corrective With Humor; Note that analyses are underpowered due to administrative issues with funding that halted recruitment early; Test type: Superiority; p = 0.008, ANCOVA — Sidak's adjusted p-value for multiple comparisons; DF = 6; Mean Difference (Final Values) = -6.469932, 95% CI 2-sided [-11.58151 to -1.358358], Standard Error of Mean 2.102231 — Humor - control

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | Vaccine Corrective Control | Vaccine Corrective With Economic Recovery Framing | Vaccine Corrective With Freedom Framing | Vaccine Corrective With Humor
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/24 | 0/22

LIMITATIONS AND CAVEATS:
Limitations include the ANCOVAs being underpowered. Failure to reject the null offers limited value because there's not strong support for lack of effect. Beliefs were also measured on a continuous scales, which can detect even small effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT05085613/Prot_SAP_000.pdf